CLINICAL TRIAL: NCT03512418
Title: Development of Ingestible Biosensors to Enhance PrEP Adherence in Substance Users (PrEPSteps)
Acronym: PrEPSteps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gilead Sciences (Industry); The Fenway Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Peter R Chai MD, Emergency Medicine Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019P000792; K23DA044874 (NIH)
Record Dates: First submitted 2018-03-21; First posted 2018-04-30 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Substance Use Disorders
Keywords: HIV Prevention; Pre-exposure Prophylaxis; Digital Pill; Substance Use Disorder
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- PrEPsteps (Experimental): Participants receive the digital pills with Truvada, plus the PrEPsteps intervention that is programmed at the randomization study visit (Study Visit 2). Participants will use PrEPsteps and the digital pill to measure Truvada adherence for months 1-3.
  Interventions: Behavioral: PrEPsteps; Device: Digital pill; Drug: Truvada
- Control (Active Comparator): Participants receive digital pills with Truvada alone. Participants will use digital pills with Truvada for months 1-3.
  Interventions: Device: Digital pill; Drug: Truvada

INTERVENTIONS:
Behavioral: PrEPsteps — Smartphone-based adherence intervention based in 1) LifeSteps, 2) Contingent Reinforcement/Corrective Feedback, and 3) Screening Brief Intervention and Referral to Treatment (SBIRT).
  Arms: PrEPsteps
Device: Digital pill — The digital pill comprises a standard gelatin capsule with an integrated radiofrequency emitter that overencapsulates the desired medication (Truvada). When participants ingest the digital pill, the chloride ion gradient in the stomach activates the radiofrequency emitter which transmits direct evidence of medication ingestion to a wearable reader which relays this data to the participant's smartphone and cloud server.
Drug: Truvada — Participants receive once daily Truvada as PrEP to prevent HIV.

SUMMARY:
This study will deploy a novel, personalized, smartphone-based intervention (PrEPSteps) that responds to real-time PrEP adherence and nonadherence detected through the use of a digital pill. The PrEPSteps intervention will be developed and refined through a series of focus groups. Participants will be screened at the Screening Visit, and, if eligible, will then begin using the digital pill system at Study Visit 1 for 2 weeks. At Study Visit 2, participants will undergo randomization to using either PrEPSteps + the digital pill, or the digital pill alone to measure PrEP adherence, for 90 days. Participants will then complete 3 monthly study visits (Study Visits 3-5) where the investigators will assess digital pill adherence, conduct manual pill counts, obtain dried blood spots to confirm adherence, provide substance use disorder counseling, and obtain urine drug screens. At Study Visit 5, the investigators will conduct a semi-structured qualitative interview with participants in the PrEPsteps arm, which will be grounded in the Technology Acceptance Model, in order to understand the user response to PrEPSteps and the digital pill. All participants will complete the final follow-up assessment 3 months after Study Visit 5 (Study Visit 6).

DETAILED DESCRIPTION:
PrEPSteps is a novel, smartphone-based behavioral intervention that delivers PrEP adherence messages in response to detected PrEP ingestion via an innovative digital pill. PrEPSteps comprises 1) an adaptation of LifeSteps, an evidence-based medication adherence behavioral intervention, with smartphone-delivered booster sessions, 2) messages of contingent reinforcement and corrective feedback, and 3) stimulant use screening, brief assessment, and referral to treatment. In this K23, the investigators will first refine and inform the specification of PrEPSteps with a series of focus groups. The investigators will next test the feasibility, acceptability and potential for an effect of PrEPSteps to boost PrEP adherence in a pilot randomized controlled trial of men who have sex with men (MSM) with stimulant use. Finally, the investigators will conduct qualitative interviews among participants who used PrEPSteps to understand the participant response to living with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender MSM
* Moderate to severe non-alcohol substance use disorder
* Self-reported missed PrEP doses (> or equal to 2 doses in 1 week over past 3 months)
* HIV negative
* On PrEP or initiating PrEP
* Has qualifying laboratory testing: Cr clearance, HBV, liver function tests
* Owns a smartphone with Android or iOS
* Age 18 or older

Exclusion Criteria:

* Non-English speaker
* HIV positive
* History of Crohn's disease or ulcerative colitis
* History of gastric bypass, bowel stricture
* History of GI malignancy or radiation to abdomen
* Unable/unwilling to ingest a digital pill
* Allergy to gelatin, silver or zinc (components of the digital pill)
* Does not qualify for PrEP (abnormal liver function, or Cr Clearance <60)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender men who have sex with men (MSM)
Enrollment: 30 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Chai, MD, MMS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Fenway Health, Boylston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chai PR, Lee JS, Goodman GR, Albrechta H, Hokayem J, Loo L, Mohamed Y, Glynn TR, Rosen RK, Mayer KH, Boyer EW, Alpert P, Buffkin E, Carnes C, O'Cleirigh C. PrEPSteps: A Pilot Randomized Controlled Trial to Assess the Feasibility and Acceptability of a Digital Pill-Based PrEP Adherence Intervention in Men Who Have Sex with Men with Substance Use Disorder. AIDS Behav. 2026 Feb 2. doi: 10.1007/s10461-026-05049-x. Online ahead of print. PMID 41627697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a health clinic in Boston, MA. We also conducted community-based outreach in the greater Boston metropolitan area through flyers and postings. Interested participants contacted the study team and were prescreened for eligibility criteria.
Pre-assignment Details: Potentially eligible participants were consented and started on the digital pill system (DPS). Standardized training was completed and participants were asked to use the DPS for 2 weeks as a run-in period prior to randomization.
Groups:
- PrEPSteps (Intervention): A text-based cognitive behavioral adherence intervention delivered in response to adherence data obtained through a digital pill system (ingestible radio frequency system co-encapsulated with tenofovir disoproxil fumarate/emtricitabine). In response to nonadherence dates detected by the digital pill, PrEPSteps sends personalized adherence interventions presenting barriers to adherence and solutions to these barriers in real-time.
- Control: Operation of the digital pill system to measure daily adherence to tenofovir disoproxil fumarate/emtricitabine. Participants were trained on the use of the digital pill system and asked to operate it daily to record adherence.
Period: Overall Study
Arm/Group | PrEPSteps (Intervention) | Control
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEPSteps (Intervention) | Control | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 38 [22 to 54] | 37.5 [25 to 59] | 37.5 [22 to 59]
Sex: Female, Male [Count of Participants; unit: Participants] — Male/female at birth
  Participants
    Female | 0 | 0 | 0
    Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 9 | 21
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Number of sexual partners [Median (Full Range); unit: partners] — number of sexual partners by self report in the past 3 months.
  partners | 14.8 [0 to 30] | 3.36 [0 to 30] | 3.5 [0 to 30]
Substance use during sex [Median (Inter-Quartile Range); unit: events] — Self reported instances of substance use before or during sex in the past 3 months. Participants self report the number of instances. The value does not indicate a better or worse outcome.
  events | 3.5 [0 to 65] | 2.5 [0 to 50] | 3 [0 to 65]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Adherence Intervention Qualitative and Quantitive Questionnaire
Description: Number of participants who were able to complete the trial and record adherence events using the digital pill system in the intervention arm.
Time Frame: three month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | PrEPsteps | Control
Number analyzed (Participants) | 14 | 14
Participants | 14 | 14

2. Secondary Outcome: Potential of PrEPsteps to Improve Adherence
Description: Number of digital pill recorded ingestions at week 13 (end of intervention period) recorded as percent adherence
Time Frame: three month study visit
Measure: Mean (Standard Deviation); unit: percentage of pills taken appropriately
Arm/Group | PrEPsteps | Control
Number analyzed (Participants) | 14 | 14
percentage of pills taken appropriately | 86 (17.23) | 72 (33.14)

3. Secondary Outcome: Number of People Who Found the Digital Pill Acceptable to Use Within the Intervention Arm
Description: Qualitative interviews asking participants if they found the use of the digital pill system acceptable and did not interfere with their daily PrEP use. This outcome was only assessed in the PrEPSteps (intervention arm) only.
Time Frame: three month visit
Population: Only intervention arm (PrEPSteps) completed qualitative interviews at the 3 month study endpoint for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEPsteps
Number analyzed (Participants) | 14
Participants | 14

4. Other Pre Specified Outcome: Accuracy of Digital Pill Compared to Pill Counts and Dried Blood Spot for Adherence
Description: Accuracy of digital pill in measuring PrEP adherence as compared to dried blood spot testing for tenofovir diphosphate
Time Frame: one and three month study visits
Reporting Status: Not Posted, anticipated posting 2027-07

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PrEPsteps | Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Our study had several limitations. First, it was conducted at a single federally qualified community health center with expertise in HIV treatment and prevention, which may differ from settings with less familiarity in prescribing PrEP or infrastructure to support PrEPSteps deployment. Second, our study population was predominantly white; other demographic groups at higher HIV risk, such as Black and Latinx individuals with potential medical mistrust, might have different perspectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03512418/Prot_SAP_002.pdf